CLINICAL TRIAL: NCT04950361
Title: Follow-up of Patients With Talocalcaneal Coalitions
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020197
Record Dates: First submitted 2021-06-25; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Talocalcaneal Coalition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: talocalcaneal coalition — patients with talocalcaneal coalition

SUMMARY:
The objective of this study was to develop a new classification system based on the articular facets involved to cover all coalitions and guide operative planning.

DETAILED DESCRIPTION:
Patients were diagnosed with talocalcaneal coalition using a CT scan, between January 2009 and February 2021. We classified the coalition into four main types according to the shape and nature of the coalition: I, inferiorly overgrown talus or superiorly overgrown calcaneus; II, both talus and calcaneus overgrew; III, coalition with an accessory ossicle; (I-III types are non-osseous coalition) IV, complete osseous coalition. Then each type was further divided into three subtypes according to the articular facets involved. A, the coalition involving the anterior facets; M, the coalition involving the middle facets, and P, the coalition involving the posterior facets.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as talocalcaneal coalition by CT or MRI at the outpatient
* Underwent arthroscopic talocalcaneal coalition resection due to failure of conservative treatment

Exclusion Criteria:

* The affected side underwent other foot and ankle operations
* Combined with other ankle diseases
* Refused to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that were diagnosed with talocalcaneal coalition using a CT scan, between January 2009 and February 2021.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
CT | pre-surgery
  computerized tomography scan

SECONDARY OUTCOMES:
MRI | pre-surgery
  magnetic resonance imaging
AFOAS | pre-surgery, one year after sugery
  he American Orthopaedic Foot & Ankle Society score
Tegner | pre-surgery, one year after sugery
  the Tegner score

CONTACTS AND LOCATIONS:
Overall Officials: Qinwei Guo, MD, Study Chair — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No